CLINICAL TRIAL: NCT05606510
Title: The Effects of Mindful Exercise on the Physical and Psychological Consequences of Older Priamry Osteoporotic Patients With Back Pain
Brief Title: The Effects of Mindful Exercise on Back Pain in Older Patients With Primary Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XW[2022]
Record Dates: First submitted 2022-10-21; First posted 2022-11-04 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Older People; Primary Osteoporosis; Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A 12-week, group-based mindful exercise program which will be conducted 5 times per week, 30 minutes per session.
  Interventions: Other: Mindful exercise
- Control (Other): Routine medicine, nursing care, and hospital-recommended exercise.
  Interventions: Other: usual care

INTERVENTIONS:
Other: Mindful exercise — In this study, a modified mindful exercise (ME) program based on mindful standing yoga refers to a type of exercise that aims to harmonize the body and mind through the effect of mindfulness meditation and stretching-awareness to carry on the actual moment through body movement and surroundings without any judgement.
  Arms: Intervention
Other: usual care — Routine medicine and nursing care; as well as hospital-recommended movements (physical stretching).
  Arms: Control

SUMMARY:
The goal of this randomized control trial is to determine the effects of a mindful exercise program on physical (back pain and balance) and psychological (mindfulness, kinesiophobia, anxiety and depression) consequences of primary osteoporosis in older patients. The main questions it aims to answer are:

* What are the levels of pain, balance, mindfulness, kinesiophobia, anxiety and depression in older patients with primary osteoporosis?
* Are there differences in pain, balance, mindfulness, kinesiophobia, anxiety and depression according to sociodemographic-clinical characteristics of the patients?
* Are there differences in pain, balance, mindfulness, kinesiophobia, anxiety and depression between the intervention (mindful exercise) and control (usual care) groups of older patients with primary osteoporosis?

  128 participants who meet the criteria will be recruited from the pain department of a Tertiary A level provincial Traditional Chinese Medicine hospital in Mainland China, and randomly assigned to the intervention group or control group. All patients in both groups will receive usual care, including routine medicine and nursing care. The study will last for 12 weeks (one-week training in hospital and 11-week on-line sessions at home) and 4-week follow up.

Patients in the intervention group will receive a group-based mindful exercise which will be conducted 5 times per week, 30 minutes per session, and co-led by a mindfulness-trained main researcher and a professional exercise specialist for the first week (week 1) hospitalization. When they discharge, on-line sessions (week 2-12) will be conducted by the main researcher from Monday to Friday. Patients and primary caregivers will be taught how to use 'Tencent meet' software. Upon discharge, a WeChat group will be set up to notify the exercise time and send the links for the online sessions. Those in the control group will received routine medicine and nursing care as usual, and only be taught on the hospital-recommended movements (physical stretching) and encouraged to do it at home on their own. All the variables (pain, mindfulness, kinesiophobia, anxiety and depression) and the TUG test (balance) will be measured at the following time point: baseline (Time 1), week 4 (Time 2), week 8 (Time 3), week 12 (Time 4, immediately post-intervention) and week 16 (Time 5, 4 weeks after the intervention) for the two groups of patients.

The study will obtain ethical clearance from the study setting, as well as written consent from the participants. Descriptive statistics will be computed for all variables. Normality and homogeneity of the variances will be tested using the Shapiro-Wilk and Levene tests, respectively. The data will be analyzed using mixed-model analysis of variance to test the main and interaction effects of group (independent factor) and time (repeated-measures factor) on the dependent variables. The findings of the study would certainly have implications for the treatment of older patients with primary osteoporosis, especially non-pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years and above, and can use smart phone.
* Patients diagnosed as primary osteoporosis with mild to moderate back pain [Numeric Rating Scale (NRS) score 1-6] for more than 3 months.
* Patients with low risk of falls that measured by the Morse Fall Risk Scale (MFS) [MFS score <25].
* Patients with no visual, hearing, mental problems or cognitive impairment [assessed using Short Portable Mental Status Questionnaire] that could prevent communication.
* Patients with no secondary diseases resulting in decreased mobility, functional status.
* Patients with no neurological or muscle diseases, ability to continuously attend the exercise program.

Exclusion Criteria:

* Patients with secondary osteoporosis or other diseases that can interfere with bone metabolism.
* Patients taking of concomitant medication that affected calcium and bone metabolism.
* Patients who presence of medical conditions that could have interfered with the outcomes of the trial.
* Patients with cardiovascular or cerebrovascular disease (blood pressure higher than 160/110 mmHg on medication, with systolic blood pressure less than 90 mmHg, with heart stents or body implantation, with a history of thrombosis within the past 6 months).
* Patients who are in the rehabilitation period for surgical intervention.
* Patients who have not recovered from muscle strain, joint injuries or fractures (fractures within the past three months).
* Patients undergoing other psychotherapy, including taking psychotropic medications.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of back pian level | 0,4,8,12,16 weeks post-intervention
  Back pain will be measured using the Chinese version of Global Pain Scale (GPS), which has 20 items with four dimensions: pain, feelings, clinical outcomes, activities. Each item is rate with 11-point scale ranging from 0-10. The total score is 0 to 200 points and the higher the score, the higher the pain intensity and interference.
Change of balance ability | 0,4,8,12,16 weeks post-intervention
  Balance will be measured by the Timed Up and Go (TUG) test using the following equipment: stopwatch, standard chair (chair with about 46 cm high and the armrest about 20 cm high), the measured distance of 3 meters (Zakaria et al., 2015). There is no official cut-off for TUG, but previous study implied that a score of >12 seconds indicates a high risk of falling.
Change of mindfulness level | 0,4,8,12,16 weeks post-intervention
  Mindfulness will be measured using the Chinese version the short form of the Five Facet Mindfulness Questionnaire (FFMQ-SF), which consists 20 items with five dimensions: Observing; Describing; Acting with-awareness; Nonjudging to inner experience; Nonreacting to inner experience. Each item is scored on a 5-point Likert-type scale ranging from 1 (never or very rarely true) to 5 (very often or always true) with a total score of 20 to 100. The higher scores indicating a high level of mindfulness.
Change of kinesiophobia level | 0,4,8,12,16 weeks post-intervention
  Kinesiophobia will be measured using the Chinese version of the Tampa Scale of Kinesiophobia-11 (TSK-11) which contains 11 items with three dimensions: Somatic focus (6 items), Activity avoidance (3 items), and Avoidance beliefs (2 items). Each item was rated on a four-point Likert scale from 1 (strongly disagree) to 4 (strongly agree). A total score ranging from 11 to 44. The higher scores correspond to a greater perceived level of kinesiophobia.

SECONDARY OUTCOMES:
Change of anxiety and depression level | 0,4,8,12,16 weeks post-intervention
  Anxiety and Depression will be measure using the Chinese version of Hospital Anxiety and Depression Scale (HADS) which has 14 items with 2 subscales of anxiety and depression. Each item is scored on 0 to 3. According to the standards of the original authors, a total score of 0 to 7 represents no anxiety or depression, 8 to 10 refers to possibly or borderline anxiety or depressiom, and 11 to 21 represents possible significant anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Fei Lyu, Principal Investigator — Yunnan University of Traditional Chinese Medicine
Locations (1):
- First Affiliated Hospital of Yunnan University of Traditional Chinese Medicine, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No